CLINICAL TRIAL: NCT07031921
Title: Ultrasound Image Bank: Advancing Medical Research and Diagnostics
Acronym: Ultra-Bank
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7692
Record Dates: First submitted 2025-05-29; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Gynecological Imaging; Ultrasound Diagnostics; Gynecologic Disease
Keywords: Ultrasound Imaging
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study titled "Ultrasound Image Bank: Advancing Medical Research and Diagnostics", sponsored by the Fondazione Policlinico Universitario A. Gemelli IRCCS, aims to create a large-scale database of gynecological ultrasound images. These images will be collected during routine clinical care from both healthy patients and those with benign or malignant gynecological conditions. The goal is to support medical training, clinical research, and the development of artificial intelligence (AI) models for diagnostic purposes.

This is a prospective, observational, single-center study, with an expected enrollment of approximately 25,000 patients over five years. The ultrasound images will be linked to histological outcomes (for those undergoing surgery within 3 months) or to follow-up scans at 1 year, to enhance early diagnosis and personalized treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* All patients examined at Class Ultrasound OMIC of Fondazione Policlinico Gemelli, IRCCS in Rome.
* All patients can be enrolled regardless the results of ultrasound examination: no evidence of disease, suspicion of benign or malignant pathologies
* Aged ≥ 18 years old
* Patients who were previously enrolled and their outcome has been completed
* Signature of informed consent

Exclusion Criteria:

* No signed informed consent;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All patients who come to undergo an ultrasound examination at the Class Ultrasound OMIC Center fulfilling the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of a digital ultrasound image biobank including follow-up data | Up to 12 months after initial ultrasound examination (including follow-up data)
  Systematic prospective collection and storage of 2D ultrasound images and video clips from patients undergoing gynecological ultrasound examinations. Each record will be associated with follow-up data, including histological results (within 3 months post-surgery, if applicable) and/or ultrasound re-evaluation (at 1-year follow-up). The goal is to generate a comprehensive image biobank for future research, including artificial intelligence studies.

SECONDARY OUTCOMES:
Percentage of enrolled patients with complete follow-up data (histological results or 1-year ultrasound) | Up to 12 months after initial ultrasound examination
  Proportion of patients for whom follow-up data are available, defined as histological examination results within 3 months for those undergoing surgery, or ultrasound follow-up findings at 1 year for those not undergoing surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Carla Testa, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy